CLINICAL TRIAL: NCT01819506
Title: Patient-Targeted Upper Extremity Rehabilitation After Stroke
Brief Title: Patient Targeted Upper Extremity Rehabilitation After Stroke
Acronym: TARG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N0799-R
Record Dates: First submitted 2013-03-11; First posted 2013-03-27 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: rehabilitation; occupational therapy; upper extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted Task Practice (Experimental): Targeted task practice is defined as a therapy program aimed at patient-specific upper extremity motor impairment levels and systematically progressed to assure an ongoing "just right" match between task-difficulty and patient-ability. Participants attended occupational therapy 3 times per week for 4 weeks. Each therapy session was 2 hours in length.
  Interventions: Behavioral: Task Practice Physical Rehabilitation Therapy
- Non-Targeted Task Practice (Active Comparator): Non-targeted task practice is a standard of care treatment consisting of task practice with no guidance from the measurement framework to systematically address specific upper extremity motor impairment levels or progress rehabilitation therapy. Participants attended occupational therapy 3 times per week for 4 weeks. Each therapy session was 2 hours in length.
  Interventions: Behavioral: Task Practice Physical Rehabilitation Therapy

INTERVENTIONS:
Behavioral: Task Practice Physical Rehabilitation Therapy — Similar to stroke rehabilitation occupational therapy.
  Other Names: Task Practice

SUMMARY:
Each year in the US, approximately 795,000 people have a stroke, and the overwhelming majority of those who survive are unable to resume meaningful daily activities because of impaired movement in one arm/hand. This study will investigate the effects of a challenging 4-week physical rehabilitation therapy program that is targeted at specific movement impairments and systematically progressed to assure an ongoing "just right" level of rigor. The investigators anticipate that therapy targeted to address specific movement impairments will improve recovery of arm/hand movement in people who have had a stroke.

DETAILED DESCRIPTION:
The overwhelming majority of individuals who survive stroke have persistent upper extremity (UE) motor deficits which interfere with re-engagement in meaningful activities. While advances from neuroscience are spurring development of new rehabilitation strategies, the development of novel measurement methods has not kept pace. Currently, there is no comprehensive measurement framework to objectively quantify impairment, match a rehabilitation therapy program to a patient's impairment level, and measure specific therapy effects. Therefore there has not been a rehabilitation trial where a measurement framework is the basis for designing the treatment as well as defining the outcome. The investigators redesigned the Fugl-Meyer UE Assessment (FMA-UE) using item response theory Rasch analysis and developed a first of its kind measurement framework that locates a patient along a continuum of impairment and directs a personalized therapy program tailored to patients' specific impairments and ability levels. The purpose of this proposed research is to empirically test this framework.

The objective of this project is to empirically test the FMA-UE measurement framework.

This study hypothesizes that therapeutic task practice at the just-right challenge of difficulty will maximize post-stroke motor skill reacquisition. It is expected that "targeted task-practice", will increase UE motor ability because task goal difficulty will be matched and systematically progressed according to patients' initial and evolving levels of ability.

This is a single-blinded study with parallel arm design, stratified sampling and blocked randomization. 120 individuals with post-stroke UE hemiparesis will be enrolled; 40 participants per 3 UE impairment levels as defined by the investigators' measurement framework. Participants will engage in 12 sessions (3x/wk for 4 weeks, 2 hrs/session) of reach-to-grasp task-practice. Within each impairment level, subjects will be randomized to a treatment group; 20 to targeted task-practice and 20 to non-targeted task-practice. Targeted task-practice is personalized to patient-specific UE motor deficits with initial targets (goals) defined according to baseline measures and targets continually progressed after every 3 therapy sessions so that the goals match the patient's evolving level of ability. Non-targeted task practice is defined as a standard of care task-practice intervention intended to increase UE use but not alter specific impairments. Data analyses will include (1) ANOVA to test the effects of targeted vs. non-targeted therapy on UE motor ability, (2) multiple regression to model the relationship between therapy and movement adaptions occurring pre- to post-rehabilitation, and (3) growth mixture modeling to define responders and non-responders.

This project is significant because there is a pressing need for a comprehensive measurement framework to guide novel interventions designed to improve post-stroke UE motor function and define their effects.

ELIGIBILITY:
Inclusion Criteria:

Individuals are eligible for this study if they have:

* experienced a stroke at least 3 months prior that has resulted in unilateral hemiparesis.
* exhibit voluntarily paretic arm shoulder flexion 30 degrees with simultaneous elbow extension 20 degrees.
* impairment with overhead reach and wrist circumduction and fine motor dexterity.
* passive range of motion in affected shoulder, elbow and wrist within 20 degrees of normal values.

Exclusion Criteria:

Individuals are not eligible for this study if they have:

* a lesion in the brainstem or cerebellum.
* another neurological disease that may impair motor skills (e.g., Parkinson's Disease).
* pain in the affected upper extremity that would limit participation in the study intervention.
* difficulty understanding and following 3-step directions.
* difficulty sitting independently without postural support.
* an orthopedic condition or impaired corrected vision that alters the kinematics of reaching.
* are unable to travel to and remain in Charleston SC for the duration of the 4-week study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L. Woodbury, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Woodbury ML, Velozo CA, Richards LG, Duncan PW, Studenski S, Lai SM. Dimensionality and construct validity of the Fugl-Meyer Assessment of the upper extremity. Arch Phys Med Rehabil. 2007 Jun;88(6):715-23. doi: 10.1016/j.apmr.2007.02.036. PMID 17532892
- [Background] Velozo CA, Woodbury ML. Translating measurement findings into rehabilitation practice: an example using Fugl-Meyer Assessment-Upper Extremity with patients following stroke. J Rehabil Res Dev. 2011;48(10):1211-22. doi: 10.1682/jrrd.2010.10.0203. PMID 22234665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from a University Stroke Rehabilitation Research Registry.
Groups:
- MATCH: MATCH is defined as a task-practice occupational therapy program targeting patient-specific upper extremity motor impairment levels and systematically progressed to assure an ongoing "just right" match between task-difficulty and patient-ability.
  Task Practice Physical Rehabilitation Therapy: Similar to stroke rehabilitation occupational therapy.
- Usual Care: Usual Care is defined as a non-targeted task practice standard of care occupational therapy program consisting of task practice with no guidance from the measurement framework to systematically address specific upper extremity motor impairment levels or progress rehabilitation therapy.
  Task Practice Physical Rehabilitation Therapy: Similar to stroke rehabilitation occupational therapy.
Period: Overall Study
Arm/Group | MATCH | Usual Care
Started | 51 | 52
Completed | 43 | 47
Not Completed | 8 | 5
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- MATCH Targeted Task Practice: Targeted task practice is defined as a therapy program aimed at patient-specific upper extremity motor impairment levels and systematically progressed to assure an ongoing "just right" match between task-difficulty and patient-ability.
  Task Practice Physical Rehabilitation Therapy: Similar to stroke rehabilitation occupational therapy.
- Usual Care: Non-Targeted Task Practice: Non-targeted task practice is a standard of care treatment consisting of task practice with no guidance from the measurement framework to systematically address specific upper extremity motor impairment levels or progress rehabilitation therapy.
  Task Practice Physical Rehabilitation Therapy: Similar to stroke rehabilitation occupational therapy.
- Total: Total of all reporting groups
Arm/Group | MATCH Targeted Task Practice | Usual Care: Non-Targeted Task Practice | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.47 (12.61) | 57.58 (13.09) | 55.53 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 31 | 27 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 14 | 32
  White | 33 | 37 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 52 | 103

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment of the Upper Extremity
Description: The Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) is a stroke rehabilitation assessment of arm/hand movement impairment. It is traditionally scored by assigning 30 items assessing voluntary arm/hand movements and 3 items assessing reflexes an ordinal rating (0=unable, 1=partial, 2=near normal), then summing the ratings to obtain a general statement of ability. Instead of this traditional scoring method, the investigators will eliminate the reflex items, thus reporting the aggregate score possible from 0/60 to 60/60 points. Higher scores indicate greater levels of arm movement ability.
Time Frame: participants will be followed for the duration of the 4-week rehabilitation treatment, an expected average of 4 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MATCH Targeted Task Practice | Usual Care: Non-Targeted Task Practice
Number analyzed (Participants) | 51 | 52
score on a scale | 4.08 (4.39) | 2.45 (4.34)
Statistical Analysis 1: Comparison: MATCH Targeted Task Practice vs Usual Care: Non-Targeted Task Practice; Test type: Superiority; p = 0.912, ANOVA

2. Primary Outcome: Wolf Motor Function Test
Description: The Wolf Motor Function Test is an assessment of arm movement function. Subjects are timed (seconds) as they complete 15 functional movements with the paretic arm. The average time required to complete an item is reported in seconds so that lower scores (quicker completion times) indicate greater functional movement skills. Post-intervention averages were compared to baseline averages so a reduction in timed averages indicates improved movement function.
Time Frame: participants will be followed for the duration of the 4-week rehabilitation treatment, an expected average of 4 weeks.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MATCH Targeted Task Practice | Usual Care: Non-Targeted Task Practice
Number analyzed (Participants) | 51 | 52
seconds | -4.81 (8.40) | -6.51 (18.85)

3. Secondary Outcome: Surface Electromyographic (sEMG) Analysis of Functional Arm Muscle Activations
Description: sEMG analysis is an objective method to study muscle coordination during functional arm movements. Subjects will be fitted with sensors on the skin placed over 8 arm/shoulder muscles on both arms. The sensors will detect the muscle activity of these muscles during functional reaching movements. sEMG data will be recorded with a 16-channel wireless Motion Labs EMG system and processed with custom ORBIS software.
Time Frame: participants will be followed for the duration of the 4-week rehabilitation treatment, an expected average of 4 weeks.
Population: Complete and accurate data for this measure is no longer available.
Arm/Group | MATCH Targeted Task Practice | Usual Care: Non-Targeted Task Practice
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: An expected average of 4 weeks
Description: All-cause Mortality was not monitored/addressed.
Arm/Group | MATCH Targeted Task Practice | Usual Care: Non-Targeted Task Practice
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/52
Other Adverse Events (participants affected / at risk) | 5/51 | 1/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MATCH Targeted Task Practice (N=51) | Usual Care: Non-Targeted Task Practice (N=52)
subsequent stroke (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MATCH Targeted Task Practice (N=51) | Usual Care: Non-Targeted Task Practice (N=52)
Fall (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Fell on bus
sick (Gastrointestinal disorders) | 3 (3) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
cardiac problems (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT01819506/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT01819506/SAP_001.pdf